CLINICAL TRIAL: NCT05180058
Title: Development and Efficiency of Atraumatic Orogastric Tube Insertion Protocol with Combination of Wrapping, Fetal Position, Breastmilk, and Sucrose
Acronym: OGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayse Sonay Turkmen, Prof.Dr (Other)
Responsible Party: Sponsor-Investigator, Ayse Sonay Turkmen, Prof.Dr, Assoc.Prof., Karamanoğlu Mehmetbey University
Organization: Karamanoğlu Mehmetbey University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: oral nasogastric tube
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2022-11

CONDITIONS: Premature; Orogastric Tube; Oral Sucrose
Keywords: Premature; orogastric tube; oral sucrose; Wrapping
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Wrapping + Breastmilk Group (Experimental): Preterm newborns will be wrapped by the researcher 10 minutes before OGT insertion. Then, 2 ml of breast milk will be given by the researcher with a sterile syringe 2 minutes before the OGT insertion to the same newborn. Breast milk will be given slowly into the mouth of the preterm newborn, on the upper part of the tongue, through an injector. Preterm newborns will be recorded with a video camera for 10 minutes before the procedure and for 5 minutes during and after the procedure. Then, using video recordings, the pain and comfort of newborns will be evaluated at the 1st minute before the procedure, at the 1st minute and 2nd minute (4 measurements) during and after the procedure.
  Interventions: Other: Wrapping + Breastmilk Group
- Wrapping + Oral Sucrose Group (Experimental): Preterm newborns will be wrapped by the researcher 10 minutes before OGT insertion. Then, 2 ml of 20% oral sucrose will be given to the same newborn by the researcher with a sterile syringe 2 minutes before OGT insertion. Oral sucrose will be slowly introduced into the mouth of the preterm newborn on the upper part of the tongue through an injector. Preterm newborns will be recorded with a video camera for 10 minutes before the procedure and for 5 minutes during and after the procedure. Then, using video recordings, the pain and comfort of newborns will be evaluated at 1 minute before the procedure, during and after the procedure at 1 minute and 2 minutes (4 measurements).
  Interventions: Other: Wrapping + Breastmilk Group
- Fetal Position + Breastmilk Group (Experimental): The fetal position will be given to the preterm newborn immediately after 2 ml of breast milk is given by the researcher 3 minutes before OGT insertion. Breast milk will be given slowly into the mouth of the preterm newborn, on the upper part of the tongue, through an injector. The preterm newborn will remain in the fetal position for 5 minutes during and after the procedure. Newborns will be recorded with a video camera before, during and after the procedure. Then, using video recordings, the pain and comfort of newborns will be evaluated at the 1st minute before the procedure, at the 1st minute and 2nd minute (4 measurements) during and after the procedure.
  Interventions: Other: Wrapping + Breastmilk Group
- Fetal Position + Oral Sucrose Group (Experimental): The fetal position will be given to the preterm newborn immediately after 2 ml of oral sucrose is given by the researcher 3 minutes before OGT insertion. Oral sucrose will be slowly injected into the mouth of the preterm newborn on the upper part of the tongue by means of an injector. At the end of the 3rd minute, the clinic nurse will insert the OGT as part of the treatment. The preterm newborn will remain in the fetal position for 5 minutes during and after the procedure.
  Interventions: Other: Wrapping + Breastmilk Group

INTERVENTIONS:
Other: Wrapping + Breastmilk Group — Interventions applied during orogastric tube insertion
  Other Names: Wrapping + Oral Sucrose Group; Fetal Position + Breastmilk Group; Fetal Position + Oral Sucrose Group

SUMMARY:
This study aimed to reduce the pain and increase comfort during the orogastric tube insertion (OGT) procedure, which is routinely applied to feed these babies at 32-34 weeks of age, in preterm newborns with a sucking reflex.In addition, this study also aimed to develop an atraumatic OGT attachment protocol by combining wrapping, fetal position, breast milk and oral sucrose combined therapy.

It was planned as a randomized double-blind and controlled experimental study to evaluate the efficacy of using In addition, this study also planned to develop the atraumatic OGT insertion procedure through combined therapy of wrapping, fetal position, breast milk, and oral sucrose. The population of the research consists of preterm babies who are treated in the Neonatal Intensive Care Unit of Selcuk University Hospital. Babies to be sampled are preterm babies who are between 32 and 34 weeks of gestation.

Preterm newborns will be randomly divided into five groups;

* Group 1: Control
* Group 2: Wrapping + breast milk (2 ml)
* Group 3: Wrapping + oral sucrose (0.2 ml/kg 20% sucrose)
* Group 4: Fetal position + breast milk (2 ml)
* Group 5: Fetal position + oral sucrose (0.2 ml/kg 20% sucrose) In the NICU, OGT insertion will be performed by the clinical nurse as part of the treatment for preterm newborns, which the clinic physician deems necessary. The clinical nurse and clinician will be responsible for OGT insertion in preterm newborns. In this study, only wrapping, fetal positioning, oral breast milk and sucrose delivery methods will be applied to preterm newborns by the researcher. In this context, the responsibility of the researcher in the study will be to apply non-pharmacological methods to preterm newborns only before OGT insertion and to evaluate the pain symptoms in preterm newborns during and after OGT insertion.

The obtained data will be evaluated in SPSS-21 package program in computer environment. Normality tests, chi-square, t test, Anova, and advanced analysis will be used when necessary in the analysis of the data. The relationship between the mean score of the scale and other variables will be evaluated by correlation regression analysis. Significance will be accepted as p<0.05.

DETAILED DESCRIPTION:
Ethical and institutional permissions were obtained before starting to collect the data. Written consent will be obtained from all parents via a voluntary consent form. Preterm newborns will be randomly selected into 5 groups.

* Group 1 (Control Group); Wrapping+breastmilk, wrapping+sucrose, fetal position+sucrose and fetal position+breastmilk methods were not applied to preterms in the routine care group. However, in order to be an ethical practice and to provide ethical standard care intervention, verbal relaxation and soft touch applications were applied by the researcher in the procedure.
* Group 2 (Wrapping + Breastmilk Group); Preterm newborns will be wrapped by the researcher 10 minutes before OGT insertion. Then, 2 ml of breast milk will be given by the researcher with a sterile syringe 2 minutes before the OGT insertion to the same newborn. Breast milk will be given slowly into the mouth of the preterm newborn, on the upper part of the tongue, through an injector. Preterm newborns will be recorded with a video camera for 10 minutes before the procedure and for 5 minutes during and after the procedure. Then, using video recordings, the pain and comfort of newborns will be evaluated at the 1st minute before the procedure, at the 1st minute and 2nd minute (4 measurements) during and after the procedure.
* Group 3 (Wrapping + Oral Sucrose Group); Preterm newborns will be wrapped by the researcher 10 minutes before OGT insertion. Then, 2 ml of 20% oral sucrose will be given to the same newborn by the researcher with a sterile syringe 2 minutes before OGT insertion. Oral sucrose will be slowly introduced into the mouth of the preterm newborn on the upper part of the tongue through an injector. Preterm newborns will be recorded with a video camera for 10 minutes before the procedure and for 5 minutes during and after the procedure. Then, using video recordings, the pain and comfort of newborns will be evaluated at 1 minute before the procedure, during and after the procedure at 1 minute and 2 minutes (4 measurements).
* Group 4 (Fetal Position + Breastmilk Group); The fetal position will be given to the preterm newborn immediately after 2 ml of breast milk is given by the researcher 3 minutes before OGT insertion. Breast milk will be given slowly into the mouth of the preterm newborn, on the upper part of the tongue, through an injector. The preterm newborn will remain in the fetal position for 5 minutes during and after the procedure. Newborns will be recorded with a video camera before, during and after the procedure. Then, using video recordings, the pain and comfort of newborns will be evaluated at the 1st minute before the procedure, at the 1st minute and 2nd minute (4 measurements) during and after the procedure.
* Group 5 (Fetal Position + Oral Sucrose Group); The fetal position will be given to the preterm newborn immediately after 2 ml of oral sucrose is given by the researcher 3 minutes before OGT insertion. Oral sucrose will be slowly injected into the mouth of the preterm newborn on the upper part of the tongue by means of an injector. At the end of the 3rd minute, the clinic nurse will insert the OGT as part of the treatment. The preterm newborn will remain in the fetal position for 5 minutes during and after the procedure.

Newborns will be recorded with a video camera before, during and after the procedure. Then, using video recordings, the pain and comfort of newborns will be evaluated at the 1st minute before the procedure, at the 1st minute and 2nd minute (4 measurements) during and after the procedure.

Hypotheses (H1) There is a significant difference between the methods applied in the OGT insertion procedure (wrapping+breastmilk, wrapping+sucrose, fetal position+sucrose and fetal position+breastmilk) in terms of heart rate in preterms.

There is a significant difference between the methods applied in the (H2) OGT insertion procedure in terms of oxygen saturation of preterms.

(H3) There is a significant difference between the methods applied in the OGT insertion procedure in terms of the estimated pain score of preterms.

(H4) There is a significant difference between the methods applied in the OGT insertion procedure in terms of the estimated distress score of preterms.

(H5) There is a significant difference between the methods applied in the OGT insertion procedure in terms of the comfort level of preterms.

(H6) There is a significant difference between the methods applied in the OGT insertion procedure in terms of the mean of preterm pain in preterms.

ELIGIBILITY:
Inclusion Criteria:

* Gestational week is between 32 and 34 weeks
* Having breast milk
* Stable health status
* Spontaneous breathing
* Being fed by an orogastric tube
* Not being exposed to a painful procedure at least half an hour before the interventions
* Not taking opioid or non-opioid analgesics

Exclusion Criteria:

* newborns who did not meet the inclusion criteria

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — premature newborns who gestational week is between 32 and 34 weeks
Enrollment: 150 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
heart rate | 5 minutes
  heart rate before, during and after the procedure (1st and 2nd min.)
oxygen saturation values | 5 minutes
  oxygen saturation values before, during and after the procedure (1st and 2nd min.)
PIPP Scale | 5 minutes
  pain scores before, during and after the procedure (1st and 2nd min.)
comfort scale score | 5 minutes
  comfort scores before, during and after the procedure (1st and 2nd min.)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - KaramanogluMehmetbeyU, Karaman, Turkey
  - Karamanoglu Mehmetbey University, Karaman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Apaydin Cirik V, Turkmen AS, Derin E, Yilmaz N. Effectiveness of an atraumatic orogastric tube insertion protocol for the combined use of swaddling, facilitated tucking, breast milk and sucrose. Int J Nurs Pract. 2024 Dec;30(6):e13293. doi: 10.1111/ijn.13293. Epub 2024 Jul 29. PMID 39075946